CLINICAL TRIAL: NCT07211464
Title: Acceptance and Commitment Therapy Plus Exercise for Older People With Chronic Low-back Pain: A Pragmatic Cluster Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20241101005
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic Low-back Pain (CLBP); Acceptance and commitment therapy (ACT); psychological flexibility; exercise; back care education
MeSH Terms: conditions — Motor Activity | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded (participants and statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-plus-exercise group (Experimental): 8-week ACT plus back exercise group
  Interventions: Behavioral: Acceptance and commitment therapy (ACT); Behavioral: back exercise
- Exercise control group (Active Comparator): 8-week back care education plus exercise group
  Interventions: Behavioral: back exercise; Behavioral: back care education

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy (ACT) — Each 1.5-hour session will consist of a 1-hour ACT intervention and 30 minutes of exercise training. The ACT group was led by a trained ACT counsellor and a trained exercise trainer.
  Arms: ACT-plus-exercise group
Behavioral: back exercise — 30-minute exercise class
Behavioral: back care education — 1-hour interactive lesson on back care
  Arms: Exercise control group

SUMMARY:
Low back pain (LBP) is the fifth-most common disorder among older adults 60 years or older. The prevalence of LBP increases with age, with the highest prevalence occurring at 85 years old. Because many older individuals face various age-related life challenges (e.g., comorbidities, financial difficulties, and bereavement), the addition of chronic LBP (CLBP) to existing stressors may worsen their physical and psychological well-being. Unfortunately, CLBP is difficult to manage and is refractory to many existing treatments. Physiotherapy treatments alone show only modest improvements in LBP or LBP-related disability. Recent research has shown that proper pain self-management is crucial to reduce pain and disability in individuals with CLBP.

Acceptance and commitment therapy (ACT), a new mindfulness-based therapy, has been suggested for chronic pain management. ACT improves an individual's psychological flexibility, by improving their openness, awareness, and acceptance of the present moment (including pain). Combining ACT and exercise classes has the potential to improve the latter treatment's efficacy. Our recent pragmatic pilot, 2-arm cluster randomised controlled trial (RCT) on 40 older adults with CLBP revealed that eight weeks of ACT plus exercise and an 8-week back care education plus exercise program (control group) were safe, feasible, and well accepted by participants in elderly community centres. Moreover, compared to the control group, the ACT-plus-exercise group showed significantly greater improvements in pain intensity, LBP-related disability, health-related quality of life (HRQOL), and psychological flexibility immediately after treatment. These promising preliminary findings indicate that a fully powered clinical trial is warranted.

DETAILED DESCRIPTION:
Building on our pilot study, we aim to conduct a pragmatic definitive cluster RCT in multiple elderly community centres to validate our findings immediately post-treatment and to explore its potential beneficial effects 3 and 6 months after treatment. Additionally, we will conduct a mediation analysis to explore potential mediation effects of psychological flexibility on the association between post-treatment changes in LBP-related disability and the corresponding changes in HRQOL in older adults with CLBP. Collectively, the project's results have the potential to help clinicians find a novel pragmatic approach to empower community-dwelling older adults to self-manage their CLBP.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* have had non-specific LBP in or near the lumbosacral spine, with or without leg pain, that lasts for at least 3 months in the last 12 months
* Average pain intensity (in the past week) ≥ 4 on a scale of 0 to 10
* must have sought some healthcare professional treatments for CLBP in the last 12 months
* have an adequate level of proficiency in Chinese
* Mini-Mental Status Examination (MMSE) scores: 23 or above

Exclusion Criteria:

* People with malignant pain or lumbar spinal stenosis, confirmed dementia, severe cognitive impairment, or serious psychiatric or psychological disorders that may hinder their study participation will be excluded
* Individuals with Mini-Mental Status Examination (MMSE) scores below 23

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity | Baseline, immediately after treatment, at the 3- and 6-month follow-ups
  Current, worst, least, and average LBP intensities in the last 24 hours will be assessed in four days within a week before each assessment using separate 11-point NPRS. The NPRS ranges from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable". The average LBP intensity over the four days will be calculated as a composite score for data analysis.

SECONDARY OUTCOMES:
Change in Pain-related disability | Baseline, immediately after treatment, and at the 3- and 6-month follow-ups
  The Chinese version of the 24-item Roland-Morris Disability Questionnaire will be used to evaluate LBP-related disability in older adults.[21] It consists of 24 yes/no items concerning LBP-related functional limitations. The number of items with "yes" answers indicates the severity of the respondent's LBP-related disability. The maximum score is 24.
Change in Psychological flexibility | Baseline, immediately after treatment, and at the 3- and 6-month follow-ups
  Participants' psychological flexibility will be measured by The 7-item Chinese version of the Acceptance and Action Questionnaire II (AAQ-II). It comprises 7 statements, which respondents rate on a 7-point scale, where 1 means "never true" and 7 means "always true". The maximum total score is 49. Higher total scores indicate less flexibility. The AAQ-II has been cross-culturally adapted and validated among Chinese adolescents and has demonstrated satisfactory internal consistency and test-retest reliability.
Change in HRQOL | Baseline, immediately after treatment, and at the 3- and 6-month follow-ups
  Participants' HRQOL will be measured by the Chinese version of the EQ-5D-5L. It comprises 5 items related to mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each item has 5 response options ("no problem", "slight problems", "moderate problems", "severe problems", and "extreme problems/unable to"). It has been found to be useful in monitoring treatments' effects on HRQOL.
Change in Psychological factors | Baseline, immediately after treatment, and at the 3- and 6-month follow-ups
  The Hong Kong Chinese version of the 21-item Depression Anxiety Stress Scales will be used to evaluate depression (7 items), anxiety (7 items), and stress (7 items) in older adults. Each item is rated on a 4-point scale ranging from 0 ("not at all") to 3 ("most of the time"). Higher scores imply more severe mental health issues. This questionnaire and its subscales have demonstrated excellent internal consistency for assessing depression, anxiety, and stress.
Change in falling risk | Baseline, immediately after treatment, and at the 3- and 6-month follow-ups
  The Timed Up and Go test will be used to assess transfer skills and walking. It can identify community-dwelling older adults at risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: at baseline, immediately after treatment, and at the 3- and 6-month follow-ups
Access Criteria: Upon reasonable request to the principal investigator
URL: https://www.polyu.edu.hk/rs/people/academic-staff/prof-arnold-wong/